CLINICAL TRIAL: NCT01894659
Title: Oral Sucrose Versus Glucose for Procedural Pain in Premature Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Danilyn Angeles, PhD, Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 5130117
Record Dates: First submitted 2013-07-01; First posted 2013-07-10 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Neonatal Procedural Pain
MeSH Terms: interventions — Sucrose; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Neonates randomized to this arm will receive the standard of practice at Loma Linda University NICU.
- 24% oral sucrose with pacifier (Experimental): Neonates randomized to this arm will receive 24% sucrose before every painful procedure on days of life 3-7 in the NICU.
  Interventions: Other: 24% oral sucrose
- 30% oral glucose with pacifier (Experimental): Neonates randomized to this arm will receive 30% oral glucose before every painful procedure on days of life 3-7.
  Interventions: Other: 30% oral glucose

INTERVENTIONS:
Other: 24% oral sucrose
  Arms: 24% oral sucrose with pacifier
Other: 30% oral glucose
  Arms: 30% oral glucose with pacifier

SUMMARY:
Premature neonates admitted to the neonatal intensive care unit (NICU) require up to several hundred procedures during their hospitalization. Many of these are tissue-damaging procedures (TDPs) that cause pain. Through our NIH funded research, we made the novel observation that exposure to a single TDP can significantly increase ATP utilization and oxidative stress, as evidenced by increased plasma levels of hypoxanthine, uric acid and malondialdehyde in neonates exposed to TDPs as compared to controls (no TDP). Because neonates are exposed to numerous TDPs, it is relevant to explore the energy costs of repeated exposures to painful procedures, an important information that is currently not known, as the effect of this cumulative metabolic dysfunction could result in potentially treatable or preventable cell injury.

Oral sucrose analgesia is frequently given to relieve procedural pain in neonates on the basis of its effect on behavioral and physiological pain scores. However, we found, through our prospective, randomized, double blind study funded by NIH, that although oral sucrose significantly reduced pain scores, its administration before a single TDP (heel lance) significantly increased ATP utilization. This is evidenced by higher plasma concentrations of hypoxanthine and uric acid in neonates given sucrose compared to control neonates (no TDP, no sucrose) or neonates just given a pacifier. These novel findings raise concern because preterm neonates have limited ATP stores and are susceptible to cell injury due to ATP depletion. In addition, it raises the relevant concern: If a single dose of oral sucrose can alter ATP metabolism, what are the effects of exposure to multiple doses of oral sucrose? More importantly, what is the effect of multiple TDPs and/or multiple oral sucrose dosages on ATP utilization, oxidative stress and cell injury? This application will also explore the effect of 30% oral glucose, another sweet solution currently used to relieve pain, on ATP metabolism.

In this study, we will test the general hypothesis that exposure to multiple TDPs and/or multiple doses of oral sucrose analgesia compared to oral glucose or standard care, alter biochemical markers of ATP utilization, oxidative stress and cell injury. We will use a prospective randomized clinical research design to test this hypothesis during days of life 3-7 of human premature neonates. Increased ATP utilization will be quantified by concentrations of hypoxanthine, xanthine and uric acid measured using HPLC. Oxidative stress will be quantified by concentrations of allantoin using gas chromatography/mass spectroscopy, and cell injury will be quantified through urinary concentration of intestinal fatty acid binding protein, an early marker of enterocyte injury. Data from this application will provide insight into the cellular and biochemical effects of repetitive and accumulated TDPs and/or multiple doses of oral sucrose. With this knowledge, we will propose and test innovative strategies that will not only decrease pain but also will prevent cell injury or cell death.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects are premature infants ≤ 34 weeks gestation and ≤ 7 days of age postnatally

Exclusion Criteria:

1. requirement for surgery
2. intraventricular hemorrhage (IVH) ≥ grade 3
3. neonates on medications such as morphine, fentanyl, versed, muscle relaxants, phenobarbital, or dilantin,
4. renal injury (plasma creatinine > 1 mg/dl,
5. severe cyanotic heart disease or severe respiratory distress,
6. known abdominal wall or intestinal anomaly or injury (NEC),
7. chromosomal anomaly and (8) facial anomaly

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2014-02; Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
We will determine the relationship between oral sucrose or glucose on urinary markers of ATP utilization, oxidative stress and cell injury compared to multiple doses of oral glucose (30%) or to control group | Day of life 3-7
  To quantify ATP utilization, we will measure urinary concentrations of Hx, Xa, UA. To quantify oxidative stress, we will measure urinary concentrations of allantoin. To quantify cell injury, we will measure urinary concentrations of intestinal fatty acid binding protein.

CONTACTS AND LOCATIONS:
Overall Officials: Danilyn Angeles, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States